CLINICAL TRIAL: NCT07400783
Title: Short Bowel Syndrome: Human Intestinal Organoids to Investigate the Different Efficacy of the GLP-2 Analogue Teduglutide in Pediatric Patients With Short Bowel Syndrome
Brief Title: TED_ORG: Study on Short Bowel Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Antonino Morabito, Surgery and Pediatric Autologous Bowel Reconstruction Rehabilitation & Regenerative Medicine, Meyer Children's Hospital IRCCS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TED_ORG
Record Dates: First submitted 2026-01-20; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Short Bowel Syndrome (SBS)
MeSH Terms: conditions — Short Bowel Syndrome | interventions — teduglutide; ALX-0600

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- teduglutide-treated organoids (Other): Human intestinal organoids derived from pediatric patients with short bowel syndrome are treated in vitro with teduglutide to assess its effects on intestinal morphology, gene and protein expression, and nutrient absorption.
  Interventions: Drug: Teduglutide (ALX-0600)
- Untreated organoids (Other): Human intestinal organoids derived from pediatric patients with short bowel syndrome are maintained in vitro without exposure to teduglutide and serve as a control group for comparison.
  Interventions: Other: No Treatment Added

INTERVENTIONS:
Drug: Teduglutide (ALX-0600) — Teduglutide is a glucagon-like peptide-2 (GLP-2) analogue. In this study, teduglutide is used in vitro on human intestinal organoids derived from pediatric patients with short bowel syndrome. The intervention is applied only to organoid cultures and is not administered directly to study participants. Teduglutide-treated organoids are compared with untreated control organoids to evaluate differences in intestinal structure, gene and protein expression, and nutrient absorption.
  Arms: teduglutide-treated organoids
Other: No Treatment Added — No Treatment Added
  Arms: Untreated organoids

SUMMARY:
The goal of this clinical trial is to understand why pediatric patients with short bowel syndrome respond differently to treatment with the glucagon-like peptide-2 (GLP-2) analogue teduglutide. Short bowel syndrome is a rare and severe condition in children that results from extensive intestinal resection and leads to impaired nutrient absorption, chronic diarrhea, and dependence on parenteral nutrition. Although teduglutide is known to promote intestinal adaptation and improve absorption, the clinical response varies widely among patients, and the biological mechanisms underlying this variability are not fully understood.

This study aims to investigate the effects of teduglutide using human intestinal organoids derived from intestinal tissue samples of pediatric patients with short bowel syndrome. Intestinal organoids are three-dimensional structures grown from patient-derived stem cells that reproduce key structural and functional characteristics of the human intestine. These organoids provide a human-based experimental model that allows the study of intestinal morphology, cellular behavior, and nutrient absorption in a controlled in vitro environment.

The main questions this study aims to answer are:

Does treatment with teduglutide improve the absorptive capacity of human intestinal organoids derived from pediatric patients with short bowel syndrome?

Are there differences in intestinal structure, cellular proliferation, and gene expression between teduglutide-treated organoids and untreated organoids?

Are specific molecular or cellular features associated with different responses to teduglutide?

Researchers will compare intestinal organoids treated with teduglutide to untreated organoids obtained from the same patients. This comparison will be used to evaluate changes in organoid morphology, expression of receptors involved in intestinal growth and absorption, activity of nutrient transporters, and overall absorptive function. The study will also explore differences between organoids derived from patients who show different clinical responses to teduglutide.

Participants in this study are pediatric patients with short bowel syndrome or patients undergoing intestinal resection surgery as part of their standard clinical care. No experimental treatment is administered directly to participants as part of this study. Intestinal tissue samples are collected only during clinically indicated surgical procedures and are not obtained specifically for research purposes.

Participants will:

Provide intestinal tissue samples collected during routine or clinically indicated intestinal surgery

Have intestinal organoids generated from their tissue samples using established laboratory techniques

Have their organoids studied in vitro with and without exposure to teduglutide to evaluate intestinal structure, gene and protein expression, and nutrient absorption mechanisms

The results of this study are expected to improve understanding of the biological mechanisms underlying variable responses to teduglutide and may contribute to the development of more personalized treatment strategies for pediatric patients with short bowel syndrome in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients or His/her Parents/ legal guardian must provide informed consent before they can participate in the study.
* Paediatric patients: Male and female patients aged ≥ 4 months old and ≤ 18 years;
* SBS patient or patient undergoing intestinal resective surgery

Exclusion Criteria:

* Adult patients (≥ 18 years old);
* Patients who have never undergone intestinal resective surgery
* Current or past use of teduglutide

Ages: 4 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Intestinal organoid diameter after in vitro exposure to teduglutide | During in vitro treatment period (up to 7 days)
  Quantitative measurement of intestinal organoid diameter assessed by image-based analysis in patient-derived human intestinal organoids treated in vitro with teduglutide and compared with untreated organoids from the same participant.
Crypt-villus-like architecture in intestinal organoids | During in vitro treatment period (up to 7 days)
  Quantitative assessment of crypt-villus-like architectural features in patient-derived human intestinal organoids following in vitro exposure to teduglutide, evaluated by image-based morphological analysis and compared with untreated organoids from the same participant.
Organoid shape (sphericity) after in vitro teduglutide treatment | During in vitro treatment period (up to 7 days)
  Quantitative measurement of organoid shape, expressed as sphericity index, in patient-derived human intestinal organoids treated in vitro with teduglutide and compared with untreated organoids from the same participant.
Lumen size in intestinal organoids after in vitro exposure to teduglutide | During in vitro treatment period (up to 7 days)
  Quantitative measurement of lumen size assessed by image-based analysis in patient-derived human intestinal organoids treated in vitro with teduglutide and compared with untreated organoids from the same participant.
Intestinal organoid volume after in vitro exposure to teduglutide | During in vitro treatment period (up to 7 days)
  Quantitative measurement of intestinal organoid volume assessed by image-based analysis in patient-derived human intestinal organoids treated in vitro with teduglutide and compared with untreated organoids from the same participant.
Lumen integrity in intestinal organoids after in vitro exposure to teduglutide | During in vitro treatment period (up to 7 days)
  Quantitative assessment of lumen integrity assessed by image-based analysis in patient-derived human intestinal organoids treated in vitro with teduglutide and compared with untreated organoids from the same participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Aou Meyer IRCSS, Florence, Florence, Italy